CLINICAL TRIAL: NCT05887375
Title: A Double-blind, Randomized, Parallel Group Study to Compare Rocuronium Reversal With Sugammadex (Bridion®) Versus Neostigmine/Glycopyrrolate and the Incidence of Urinary Retention After Elective Ambulatory Posterior Lumbar Laminectomy
Brief Title: Sugammadex vs Neostigmine/Glycopyrrolate on Urinary Retention After Spine Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Julie Marshall, Professor of Anesthesiology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2096001; MISP Database number 101357 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-04-25; First posted 2023-06-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Spine Surgery; Reversal of Neuromuscular Blockade; Urinary Retention Postoperative
Keywords: Urinary retention; Spine surgery; Sugammadex; Neostigmine; Neuromuscular blockade; Neuromuscular blockade reversal; Cholinesterase Inhibitors; Cholinergic Agents; Physiological Effects of Drugs; Parasympathomimetic; Autonomic Agents
MeSH Terms: conditions — Urinary Retention | interventions — Sugammadex; Neostigmine; Glycopyrrolate; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex 2 mg/kg (Experimental): Sugammadex 2 mg/kg administered as a single intravenous (IV) dose.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Neostigmine + Glycopyrrolate (Active Comparator): Neostigmine 50 μg/kg (up to 5 mg maximum dose) plus glycopyrrolate 10 μg/kg (up to 1 mg maximum dose) administered as a single IV dose.
  Interventions: Drug: Neostigmine; Drug: Glycopyrrolate; Drug: Rocuronium

INTERVENTIONS:
Drug: Sugammadex — Sugammadex will be used to reverse rocuronium neuromuscular blockade (NMB). Dose will be according to participant actual body weight.
  Other Names: Bridion; MK-8616
  Arms: Sugammadex 2 mg/kg
Drug: Neostigmine — Neostigmine will be used to reverse rocuronium NMB. Dose will be according to participant actual body weight.
  Other Names: Bloxiverz
  Arms: Neostigmine + Glycopyrrolate
Drug: Glycopyrrolate — Glycopyrrolate will be co-administered with neostigmine during reversal of rocuronium NMB. Dose will be according to participant actual body weight.
  Other Names: Glycopyrrolate injection, USP
  Arms: Neostigmine + Glycopyrrolate
Drug: Rocuronium — To achieve NMB, participants will receive the steroidal neuromuscular blocking agent Rocuronium Bromide administered via IV infusion and dosed according to participant actual body weight. It will be used per label to maintain muscle relaxation as an adjunct to general anesthesia.
  Other Names: Rocuronium Bromide

SUMMARY:
This is an active-comparator controlled study to evaluate the effect of sugammadex compared to neostigmine/glycopyrrolate for reversal of rocuronium on the incidence of urinary retention after subjects undergo elective ambulatory spine surgery.

DETAILED DESCRIPTION:
Subjects requiring elective ambulatory posterior lumbar laminectomy, will receive either an intravenous infusion bolus of Sugammadex (2 mg/kg dosed by actual body weight) or intravenous infusion bolus of Neostigmine (50 μg/kg, up to 5 mg maximum dose) plus Glycopyrrolate (10 μg/kg, up to 1 mg maximum dose). Additionally, all subjects will receive hospital standard of care therapy for their surgery and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA Physical Status I-III

Exclusion Criteria:

* Inability to obtain written informed consent
* Allergy to medications used in the protocol
* Known or suspected neuromuscular disorders
* Significant renal disease with a serum creatinine ≥ 2 mg/dL
* Significant liver disease
* A family history of malignant hyperthermia
* History of genitourinary surgery, cancer, or radiation within the last year
* Currently prescribed urological medications or diuretics
* BPH or symptoms of BPH (interrupted or weak urine stream or wake up to urinate more than two times per night)
* History or diagnosis of urinary incontinence or urinary retention
* History of PONV with use of scopolamine
* Use of Foley catheter pre- or intra- operatively
* Perioperative medications that influence micturition (e.g., diuretics or intraoperative anticholinergic medication use other than NMB reversal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of urinary retention | Up to 6 hours after administration of study intervention
  The difference between sugammadex and neostigmine/glycopyrrolate on the incidence of urinary retention defined as no void more than 6 hours after posterior lumbar spine surgery in ambulatory/short stay patients.

SECONDARY OUTCOMES:
Micturition | Up to 1 day after administration of study intervention
  Between patients who received sugammadex and neostigmine/glycopyrrolate. To compare actual times of micturition we will analyze the proportion of patients (percentages) voided at 6, 9, 12 and 24 hours.
Bladder urine volume | Up to 6 hours after administration of study intervention
  Between patients who received sugammadex and neostigmine/glycopyrrolate. To compare bladder urine volumes in milliliters (mL) we will perform bladder ultrasound scan at 6 hours postoperatively if patients did not void.
Urinary retention symptoms | Up to 1 day after administration of study intervention
  Between patients who received sugammadex and neostigmine/glycopyrrolate. To compare urinary retention symptoms, we will administer a questionnaire at 6 hours postoperatively and on postoperative day 1.
Bladder catheterization | Up to 1 Day after administration of study intervention
  Between patients who received sugammadex and neostigmine/glycopyrrolate. To compare need for bladder catheterization (straight or Foley).
Length of hospital stay | Up to 7 Days after administration of study intervention
  Between patients who received sugammadex and neostigmine/glycopyrrolate. To compare length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Mraovic, MD, FASA, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldini G, Bagry H, Aprikian A, Carli F. Postoperative urinary retention: anesthetic and perioperative considerations. Anesthesiology. 2009 May;110(5):1139-57. doi: 10.1097/ALN.0b013e31819f7aea. PMID 19352147
- [Background] McLain RF, Kalfas I, Bell GR, Tetzlaff JE, Yoon HJ, Rana M. Comparison of spinal and general anesthesia in lumbar laminectomy surgery: a case-controlled analysis of 400 patients. J Neurosurg Spine. 2005 Jan;2(1):17-22. doi: 10.3171/spi.2005.2.1.0017. PMID 15658121
- [Background] Chang Y, Chi KY, Tai TW, Cheng YS, Lee PH, Huang CC, Lee JS. Risk factors for postoperative urinary retention following elective spine surgery: a meta-analysis. Spine J. 2021 Nov;21(11):1802-1811. doi: 10.1016/j.spinee.2021.05.009. Epub 2021 May 18. PMID 34015508
- [Background] Cremins M, Vellanky S, McCann G, Mancini M, Sanzari L, Yannopoulos A. Considering healthcare value and associated risk factors with postoperative urinary retention after elective laminectomy. Spine J. 2020 May;20(5):701-707. doi: 10.1016/j.spinee.2020.01.012. Epub 2020 Jan 29. PMID 32006710
- [Background] Cha JE, Park SW, Choi YI, et al. Sugammadex use can decrease the incidence of post-operative urinary retention by avoiding anticholinergics: a retrospective study. Anesthesia and Pain Medicine. 2018;13(1):40-46.
- [Background] Zakaria HM, Lipphardt M, Bazydlo M, Xiao S, Schultz L, Chedid M, Abdulhak M, Schwalb JM, Nerenz D, Easton R, Chang V; MSSIC Investigators. The Preoperative Risks and Two-Year Sequelae of Postoperative Urinary Retention: Analysis of the Michigan Spine Surgery Improvement Collaborative (MSSIC). World Neurosurg. 2020 Jan;133:e619-e626. doi: 10.1016/j.wneu.2019.09.107. Epub 2019 Sep 27. PMID 31568914